CLINICAL TRIAL: NCT03537508
Title: A Phase III, Partially Modified Double-blind, Randomized, Parallel-group, Active-controlled, Multi-center Study to Compare the Immunogenicity and Describe the Safety of MenACYW Conjugate Vaccine and MENVEO® When Administered Concomitantly With Routine Pediatric Vaccines to Healthy Infants and Toddlers in the United States
Brief Title: Immunogenicity and Safety of a Quadrivalent Meningococcal Conjugate Vaccine When Administered Concomitantly With Routine Pediatric Vaccines in Healthy Infants and Toddlers in the US
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MET42; U1111-1183-6361 (Registry Identifier: ICTRP); 2018-001473-24 (EudraCT Number)
Record Dates: First submitted 2018-05-15; First posted 2018-05-25 (Actual); Results first posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Healthy Volunteers (Meningococcal Infection)
Keywords: Meningococcal meningitis; MenACYW conjugate vaccine; Quadrivalent meningococcal vaccine
MeSH Terms: conditions — Meningococcal Infections; Meningitis, Meningococcal | interventions — Meningococcal Vaccines; pentacel; 13-valent pneumococcal vaccine; RotaTeq; Hepatitis B Vaccines; Engerix-B; Measles-Mumps-Rubella Vaccine; Chickenpox Vaccine; Hepatitis A Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The study was conducted modified double blind for the infant part of the study, with everyone involved in the study (participants/parents, investigators, safety outcome assessor, Sponsor) blinded to the meningococcal vaccine received, except the personnel administering the vaccine.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Group 1a (Experimental): MenACYW conjugate vaccine and routine vaccines at 2, 4, 6, and 12 to 15 months of age
  Interventions: Biological: MenACYW conjugate vaccine; Biological: DTaP-IPV//Hib vaccine; Biological: Pneumococcal 13-valent conjugate vaccine; Biological: Pentavalent rotavirus vaccine; Biological: Hepatitis B vaccine; Biological: Measles, mumps, rubella (MMR) vaccine; Biological: Varicella vaccine
- Group 1b (Experimental): MenACYW conjugate vaccine at 2, 4, 6, and 15 to 18 months of age and routine vaccines at 2, 4, 6, 12 to 15 months of age, and 15 to 18 months of age
  Interventions: Biological: MenACYW conjugate vaccine; Biological: DTaP-IPV//Hib vaccine; Biological: Pneumococcal 13-valent conjugate vaccine; Biological: Pentavalent rotavirus vaccine; Biological: Hepatitis B vaccine; Biological: Measles, mumps, rubella (MMR) vaccine; Biological: Varicella vaccine; Biological: Hepatitis A vaccine
- Group 2a (Active Comparator): MENVEO® at 2, 4, 6, and 12 months of age and routine vaccines at 2, 4, 6, 12, and 15 to 18 months of age
  Interventions: Biological: MenACYW-135 conjugate vaccine; Biological: DTaP-IPV//Hib vaccine; Biological: Pneumococcal 13-valent conjugate vaccine; Biological: Pentavalent rotavirus vaccine; Biological: Hepatitis B vaccine; Biological: Measles, mumps, rubella (MMR) vaccine; Biological: Varicella vaccine
- Group 2b (Active Comparator): MENVEO® at 2, 4, 6, and 12 months of age and routine vaccines at 2, 4, 6, 12, and 15 to 18 months of age
  Interventions: Biological: MenACYW-135 conjugate vaccine; Biological: DTaP-IPV//Hib vaccine; Biological: Pneumococcal 13-valent conjugate vaccine; Biological: Pentavalent rotavirus vaccine; Biological: Hepatitis B vaccine; Biological: Measles, mumps, rubella (MMR) vaccine; Biological: Varicella vaccine; Biological: Hepatitis A vaccine

INTERVENTIONS:
Biological: MenACYW conjugate vaccine — Meningococcal polysaccharide (serogroups A, C, Y, and W) tetanus toxoid conjugate vaccine 0.5 mL, intramuscular
  Arms: Group 1a; Group 1b
Biological: MenACYW-135 conjugate vaccine — Meningococcal (Groups A, C, Y and W-135) oligosaccharide diphtheria CRM197 conjugate vaccine, 0.5 mL, intramuscular
  Other Names: MENVEO®
  Arms: Group 2a; Group 2b
Biological: DTaP-IPV//Hib vaccine — DTaP-IPV//Hib vaccine at 2, 4, 6 and 12 to 15 (Group 1a)/15-18 (Group 1b and Group 2) months of age Intramuscular
  Other Names: Pentacel®
Biological: Pneumococcal 13-valent conjugate vaccine — Pneumococcal vaccine at 2, 4, 6, and 12 months of age, Intramuscular
  Other Names: PREVNAR 13®
Biological: Pentavalent rotavirus vaccine — Rotavirus vaccine at 2, 4, and 6 months of age, oral solution
  Other Names: RotaTeq®
Biological: Hepatitis B vaccine — Hepatitis B vaccine at 2 and 6 months of age, Intramuscular
  Other Names: ENGERIX-B®
Biological: Measles, mumps, rubella (MMR) vaccine — MMR vaccine at 12 months of age, Subcutaneous
  Other Names: M-M-R® II
Biological: Varicella vaccine — Varicella vaccine at 12 months of age
  Other Names: VARIVAX®
Biological: Hepatitis A vaccine — Hepatitis A vaccine at 15 to 18 months of age
  Other Names: HAVRIX®
  Arms: Group 1b; Group 2b

SUMMARY:
The purpose of this study was to compare the immunogenicity and describe the safety of MenACYW conjugate vaccine and MENVEO® when both are administered concomitantly with routine pediatric vaccines to healthy infants and toddlers in the US.

DETAILED DESCRIPTION:
The duration of each subject's participation in the trial was approximately 16 to 19 months (Subgroup 1a) and 19 to 22 months (Subgroup 1b and Group 2), which included a safety follow up contact at 6 months after the last vaccinations.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 42 to ≤ 89 days on the day of the first study visit.
* Healthy infants as determined by medical history, physical examination, and judgment of the investigator
* Informed consent form has been signed and dated by the parent(s) or guardian, and an independent witness, if required by local regulations
* Participant and parent/guardian were able to attend all scheduled visits and to comply with all trial procedures.
* Infants who received the first dose of hepatitis B vaccine at least 28 days before the first study visit

Exclusion Criteria:

* Participation at the time of study enrollment or in the 4 weeks preceding the first trial vaccination or planned participation during the present trial period in another clinical trial investigating a vaccine, drug, medical device, or medical procedure
* Receipt of any vaccine in the 4 weeks preceding the first trial vaccination or planned receipt of any vaccine in the 4 weeks before and/or following any trial vaccination except for influenza vaccination, which could have been received at a gap of at least 2 weeks before or 2 weeks after any study vaccination. This exception included monovalent pandemic influenza vaccines and multivalent influenza vaccines
* Previous vaccination against meningococcal disease with either the trial vaccine or another vaccine (i.e., mono- or polyvalent, PS, or conjugate meningococcal vaccine containing serogroups A, C, Y, or W; or meningococcal B serogroup-containing vaccine).
* Previous vaccination against diphtheria, tetanus, pertussis, poliomyelitis, hepatitis A, measles, mumps, rubella, varicella; and of Haemophilus influenzae type b, Streptococcus pneumoniae, and /or rotavirus infection or disease
* Receipt of more than 1 previous dose of hepatitis B vaccine
* Receipt of immune globulins, blood, or blood-derived products since birth
* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy, such as anti-cancer chemotherapy or radiation therapy; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks) since birth
* Family history of congenital or hereditary immunodeficiency, until the immune competence of the potential vaccine recipient is demonstrated
* Individuals with blood dyscrasias, leukemia, lymphoma of any type, or other malignant neoplasms affecting the bone marrow or lymphatic systems
* Individuals with active tuberculosis
* History of any Neisseria meningitidis infection, confirmed either clinically, serologically, or microbiologically
* History of diphtheria, tetanus, pertussis, poliomyelitis, hepatitis B, hepatitis A, measles, mumps, rubella, varicella; and of Haemophilus influenzae type b, Streptococcus pneumoniae, and /or rotavirus infection or disease
* At high risk for meningococcal infection during the trial (specifically, but not limited to, subjects with persistent complement deficiency, with anatomic or functional asplenia, or subjects travelling to countries with high endemic or epidemic disease)
* History of intussusception
* History of any neurologic disorders, including any seizures and progressive neurologic disorders
* History of Guillain-Barré syndrome
* Known systemic hypersensitivity to any of the vaccine components or to latex, or history of a life-threatening reaction to the vaccine(s) used in the trial or to a vaccine containing any of the same substances, including neomycin, gelatin, and yeast
* Verbal report of thrombocytopenia contraindicating intramuscular vaccination in the investigator's opinion
* Bleeding disorder, or receipt of anticoagulants in the 3 weeks preceding inclusion, contraindicating intramuscular vaccination in the investigator's opinion
* Receipt of oral or injectable antibiotic therapy within 72 hours prior to the first blood draw
* Chronic illness (including, but not limited to, cardiac disorders, congenital heart disease, chronic lung disease, renal disorders, auto-immune disorders, diabetes, psychomotor diseases, and known congenital or genetic diseases) that in the opinion of the investigator, was at a stage where it might have interfered with trial conduct or completion
* Any condition which, in the opinion of the investigator, might have interfered with the evaluation of the study objectives
* Moderate or severe acute illness/infection (according to investigator judgment) on the day of vaccination or febrile illness (temperature ≥ 38.0°C [≥ 100.4°F]). A prospective participant was not included in the study until the condition has been resolved or the febrile event has been subsided
* Identified as a natural or adopted child of the investigator or employee with direct involvement in the proposed study
* The above information was not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 42 Days to 89 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2627 (Actual)
Dates: Start 2018-04-25 (Actual); Primary Completion 2023-09-22 (Actual); Study Completion 2023-09-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur, a Sanofi Company
Locations (70):
- United States (65):
  - Birmingham Pediatric Associates Site Number : 8400026, Birmingham, Alabama
  - Southeastern Pediatric Associates Site Number : 8400003, Dothan, Alabama
  - MedPharmics, LLC - Phoenix Site Number : 8400083, Phoenix, Arizona
  - Northwest Arkansas Pediatric Clinic Site Number : 8400011, Fayetteville, Arkansas
  - The Children's Clinic of Jonesboro, PA Site Number : 8400032, Jonesboro, Arkansas
  - Emmaus Research Center, Inc Site Number : 8400031, Anaheim, California
  - Premier Health Research Center Site Number : 8400007, Downey, California
  - Joint Clinical Trials Huntington Park Site Number : 8400126, Huntington Park, California
  - United Clinical Research Site Number : 8400092, Huntington Park, California
  - Matrix Clinical Research Site Number : 8400095, Los Angeles, California
  - Center for Clinical Trials, LLC Site Number : 8400030, Paramount, California
  - Center for Clinical Trials of San Gabriel Site Number : 8400076, West Covina, California
  - Asclepes Research Centers Site Number : 8400064, Brooksville, Florida
  - Avail Clinical Research Site Number : 8400077, DeLand, Florida
  - Next Phase Research Alliance Site Number : 8400057, Hialeah, Florida
  - Homestead Medical Clinic, P.A. Site Number : 8400014, Homestead, Florida
  - Next Phase Research Alliance Site Number : 8400040, Homestead, Florida
  - Children's Research, LLC Site Number : 8400063, Lake Mary, Florida
  - Axcess Medical Research Site Number : 8400068, Loxahatchee Groves, Florida
  - Acevedo Clinical Research Associates Site Number : 8400001, Miami, Florida
  - Florida Hospital Medical Group Pediatrics Site Number : 8400108, Orlando, Florida
  - IMIC Inc Site Number : 8400022, Palmetto Bay, Florida
  - Jedidiah Clinical Research Site Number : 8400132, Tampa, Florida
  - Baybol Research Institute Site Number : 8400008, Chamblee, Georgia
  - Snake River Research, PLLC Site Number : 8400073, Idaho Falls, Idaho
  - Qualmedica Research, LLC Site Number : 8400106, Evansville, Indiana
  - Brownsboro Park Pediatrics Site Number : 8400010, Louisville, Kentucky
  - All Children Pediatrics Site Number : 8400043, Louisville, Kentucky
  - ACC Pediatric Reasearch Site Number : 8400023, Haughton, Louisiana
  - Velocity Clinical Research Site Number : 8400025, Metairie, Louisiana
  - LSUHSC-Shreveport Site Number : 8400120, Shreveport, Louisiana
  - University of Maryland at The Pediatric Center of Frederick Site Number : 8400004, Frederick, Maryland
  - Virgo-Carter Pediatrics Site Number : 8400041, Silver Spring, Maryland
  - MedPharmics Biloxi Site Number : 8400080, Biloxi, Mississippi
  - Craig Spiegel, MD Site Number : 8400037, Bridgeton, Missouri
  - Creighton University Site Number : 8400039, Omaha, Nebraska
  - Tiga Pediatrics Site Number : 8400137, New York, New York
  - Blue Pediatric & Adolescent Medicine Group Site Number : 8400100, Boone, North Carolina
  - Ohio Pediatric Research Site Number : 8400084, Dayton, Ohio
  - PriMed Clinical Research Site Number : 8400002, Dayton, Ohio
  - Cyn3rgy Research Site Number : 8400085, Gresham, Oregon
  - Allegheny Health and Wellness Pavilion Site Number : 8400047, Erie, Pennsylvania
  - Coastal Pediatric Research Charleston Site Number : 8400005, Charleston, South Carolina
  - Tribe Clinical Research Site Number : 8400110, Greenville, South Carolina
  - Parkside Pediatrics - Simpsonville Site Number : 8400113, Simpsonville, South Carolina
  - Pediatric Clinical Trials Tullahoma Site Number : 8400033, Tullahoma, Tennessee
  - ARC Clinical Research at Wilson Parke Site Number : 8400059, Austin, Texas
  - Oak Cliff Research Company, LLC Site Number : 8400065, Dallas, Texas
  - Helios Clinical research Site Number : 8400075, Fort Worth, Texas
  - University of North Texas Site Number : 8400079, Fort Worth, Texas
  - University of Texas Medical Board Site Number : 8400067, Galveston, Texas
  - Helios Clinical Research Site Number : 8400109, Houston, Texas
  - Clinical Trial Network - 7080 Southwest Fwy Site Number : 8400114, Houston, Texas
  - FMC SCIENCE Site Number : 8400053, Lampasas, Texas
  - Tekton Research, Inc Site Number : 8400049, San Antonio, Texas
  - Tekton Research Site Number : 8400128, San Antonio, Texas
  - Ericksen Research and Development Site Number : 8400016, Clinton, Utah
  - Wee Care Pediatrics Site Number : 8400035, Kaysville, Utah
  - Tanner Clinic Site Number : 8400018, Layton, Utah
  - Pediatric Care Site Number : 8400056, Provo, Utah
  - Wee Care Pediatrics Roy Site Number : 8400029, Roy, Utah
  - Copperview Medical Center Site Number : 8400038, South Jordan, Utah
  - Wee Care Pediatrics Syracuse Site Number : 8400024, Syracuse, Utah
  - Alliance for Multispecialty Research Syracuse Site Number : 8400036, Syracuse, Utah
  - Marshall Health Site Number : 8400062, Huntington, West Virginia
- Puerto Rico (5):
  - Investigational Site Number : 6300116, Caguas
  - Investigational Site Number : 6300122, Guayama
  - Investigational Site Number : 6300015, San Juan
  - Investigational Site Number : 6300117, San Juan
  - Investigational Site Number : 6300140, San Juan

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Campbell JD, Gupta S, Dhingra MS, Zambrano B, Gan L, B'Chir S, Chaix J, Syrkina O, Masson J, Liabis O, Rehm C. A Phase 3 study to assess the safety and immunogenicity of a quadrivalent meningococcal conjugate vaccine (MenACYW-TT) co-administered with routine pediatric vaccines in healthy infants in the USA and Puerto Rico. Hum Vaccin Immunother. 2025 Dec;21(1):2588874. doi: 10.1080/21645515.2025.2588874. Epub 2025 Dec 3. PMID 41337697

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 69 investigational sites in Puerto Rico and the United States. Healthy infants aged >=42 to <=89 days were randomized in 2:1 ratio to either Group 1: Meningococcal polysaccharide (serogroups A, C, Y, and W) tetanus toxoid conjugate vaccine (MenACYW conjugate vaccine) and routine pediatric vaccines or Group 2: Meningococcal (groups A, C, Y, and W-135) oligosaccharide diphtheria cross reacting material (CRM) 197 conjugate vaccine (MENVEO®) and routine pediatric vaccines.
Pre-assignment Details: Each group was further divided into 2 subgroups based on the time of analyses conducted in the 2nd year of life (30 days after the 12-month vaccinations [Groups 1a and 2a] or 30 days after the 15-month vaccinations [Groups 1b and 2b], respectively. The division of the subgroups did not determine when participants received their vaccinations in the 2nd year of life. A total of 2627 participants were enrolled in this study.
Groups:
- Group 1: MenACYW Conjugate Vaccine: Participants received MenACYW conjugate vaccine 0.5 milliliter (mL) as an intramuscular (IM) injection at 2, 4, 6, and 12 to 15/15 to 18 months of age along with Pentacel® (diphtheria-tetanus-acellular pertussis [DTaP-IPV/Hib] vaccine) at 2, 4, 6 and 15 to 18 months of age; PREVNAR 13® (pneumococcal 13-valent conjugate vaccine [PCV13] at 2, 4, 6, and 12 to 15 months of age; RotaTeq® (pentavalent rotavirus vaccine [RV5]) at 2, 4, and 6 months of age; ENGERIX-B® (hepatitis B vaccine) at 2 and 6 months of age; M-M-R® II (measles, mumps, and rubella vaccine) and VARIVAX® (varicella vaccine) at 12 to 15 months of age. Additionally, participants received first dose of HAVRIX® (hepatitis A vaccine) at 15 to 18 months of age as a part of the study.
  Group 1 was divided as Groups 1a and 1b based on the time of analyses, i.e. 30 days after 12 months and 30 days after 15 months respectively. The division of the subgroups did not determine when participants received their vaccinations in the 2nd year of life.
- Group 2: MENVEO: Participants received MENVEO conjugate vaccine 0.5 mL as an IM injection at 2, 4, 6, and 12 months of age along with Pentacel (DTaP-IPV/Hib vaccine) at 2, 4, 6 and 15 to 18 months of age; PREVNAR 13 (PCV13) at 2, 4, 6, and 12 months of age; RotaTeq (rotavirus vaccine) at 2, 4, and 6 months of age; ENGERIX-B (hepatitis B vaccine) at 2 and 6 months of age; M-M-R II (measles, mumps, and rubella vaccine) and VARIVAX (varicella vaccine) at 12 months of age. In addition, they also received first dose of HAVRIX (hepatitis A vaccine) at 15 to 18 months of age.
  Group 2 was further divided as Groups 2a and 2b based on the time of analyses, i.e. 30 days after 12 months and 30 days after 15 months respectively. The division of the subgroups did not determine when participants received their vaccinations in the 2nd year of life.
Period: Overall Study
Arm/Group | Group 1: MenACYW Conjugate Vaccine | Group 2: MENVEO
Started | 1746 | 881
Safety Analysis Set (SafAS) | 1727 | 867
Vaccinated at 2 Months | 1727 | 869
Vaccinated at 4 Months | 1619 | 828
Vaccinated at 6 Months | 1543 | 793
Vaccinated at 12 Months | 1411 | 708
Vaccinated at 15 Months | 445 | 644
Completed | 1330 | 623
Not Completed | 416 | 258
Not completed — Adverse Event | 2 | 1
Not completed — Protocol Violation | 65 | 48
Not completed — Lost to Follow-up | 86 | 60
Not completed — Withdrawal by parent/guardian | 263 | 149

BASELINE CHARACTERISTICS:
Population: Baseline characteristics were assessed for all randomized participants.
Groups:
- Group 1: MenACYW Conjugate Vaccine: Participants received MenACYW conjugate vaccine 0.5 mL as an IM injection at 2, 4, 6, and 12 to 15/15 to 18 months of age along with Pentacel (diphtheria-tetanus-acellular pertussis [DTaP-IPV/Hib] vaccine) at 2, 4, 6 and 15 to 18 months of age; PREVNAR 13 (pneumococcal 13-valent conjugate vaccine [PCV13] at 2, 4, 6, and 12 to 15 months of age; RotaTeq (pentavalent rotavirus vaccine [RV5]) at 2, 4, and 6 months of age; ENGERIX-B (hepatitis B vaccine) at 2 and 6 months of age; M-M-R II (measles, mumps, and rubella vaccine) and VARIVAX (varicella vaccine) at 12 to 15 months of age. Additionally, participants received first dose of HAVRIX (hepatitis A vaccine) at 15 to 18 months of age as a part of the study.
  Group 1 was divided as Groups 1a and 1b based on the time of analyses, i.e. 30 days after 12 months and 30 days after 15 months respectively. The division of the subgroups did not determine when participants received their vaccinations in the 2nd year of life.
- Total: Total of all reporting groups
Arm/Group | Group 1: MenACYW Conjugate Vaccine | Group 2: MENVEO | Total
Number analyzed (Participants) | 1746 | 881 | 2627
Age, Continuous [Mean (Standard Deviation); unit: days] | 65.3 (8.02) | 65.3 (7.81) | 65.3 (7.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 828 | 415 | 1243
  Male | 918 | 466 | 1384
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 11 | 3 | 14
  Asian | 15 | 10 | 25
  Native Hawaiian or Other Pacific Islander | 7 | 6 | 13
  Black or African American | 204 | 99 | 303
  White | 1428 | 722 | 2150
  More than one race | 44 | 30 | 74
  Unknown or Not Reported | 37 | 11 | 48

OUTCOME MEASURES:

1. Primary Outcome: Groups 1a and 2a: Percentage of Participants With Vaccine Seroresponse Measured by Serum Bactericidal Assay Using Human Complement (hSBA) at Day 30 Post 12-Month Vaccination
Description: Functional meningococcal antibody activity against serogroups A, C, Y, and W were measured in a serum bactericidal assay utilizing the hSBA. Vaccine seroresponse was defined as a post 4th dose (Day 30 after 12-month) hSBA titer >=1:16 for participants with pre 1st dose (Day 0 before 2-month) hSBA titer less than (<) 1:8, or at least a 4-fold increase in hSBA titer from pre-vaccination to post-vaccination for participants with pre-vaccination hSBA titer >=1:8. Percentages are rounded off to the tenth decimal place.
Time Frame: Day 30 post 12-month vaccination (Month 13)
Population: Per-Protocol Analysis Set 3 (PPAS3) (for 2nd year of life vaccination). PPAS3 included participants of Full Analysis set 3 (FAS3: a subset of all randomized participants who received >=1 dose of the study vaccine in the 2nd year of life [>=12 months of age] and had a valid post-vaccination serology result in the 2nd year of life) with no relevant protocol deviations. Only those participants with data collected for each specific serogroup are reported.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Group 1a:MenACYW Conjugate Vaccine (Post 12-month Vaccination): Participants received MenACYW conjugate vaccine and routine vaccines at 2, 4, 6, and 12 to 15 months of age. The time of analyses as well as the collection of blood samples conducted in the 2nd year of life for this subgroup was 30 days after the 12-month vaccination.
- Group 2a: MENVEO (Post 12-month Vaccination): Participants received MENVEO at 2, 4, 6, and 12 months of age and routine vaccines at 2, 4, 6, 12, and 15 to 18 months of age. The time of analyses as well as the collection of blood samples conducted in the 2nd year of life for this subgroup was 30 days after the 12-month vaccination.
Arm/Group | Group 1a:MenACYW Conjugate Vaccine (Post 12-month Vaccination) | Group 2a: MENVEO (Post 12-month Vaccination)
Number analyzed (Participants) | 540 | 250
percentage of participants
  Serogroup A: number analyzed (Participants) | 501 | 223
  Serogroup A | 79.4 [75.6 to 82.9] | 77.6 [71.5 to 82.9]
  Serogroup C: number analyzed (Participants) | 530 | 238
  Serogroup C | 97.0 [95.1 to 98.3] | 88.2 [83.4 to 92.0]
  Serogroup Y: number analyzed (Participants) | 523 | 233
  Serogroup Y | 96.4 [94.4 to 97.8] | 92.3 [88.1 to 95.4]
  Serogroup W | 97.6 [95.9 to 98.7] | 96.4 [93.3 to 98.3]
Statistical Analysis 1: Comparison: Group 1a:MenACYW Conjugate Vaccine (Post 12-month Vaccination) vs Group 2a: MENVEO (Post 12-month Vaccination); Statistical analysis for Serogroup A; Test type: Non-Inferiority — The overall non-inferiority was demonstrated if the lower limit of the 2-sided 95% confidence interval (CI) was >-10% for all 4 serogroups. 95% CI of the difference was calculated from the Wilson Score method without continuity correction; Difference in Percentage of Participants = 1.86, 95% CI 2-sided [-4.38 to 8.64]
Statistical Analysis 2: Comparison: Group 1a:MenACYW Conjugate Vaccine (Post 12-month Vaccination) vs Group 2a: MENVEO (Post 12-month Vaccination); Statistical analysis for Serogroup C; Test type: Non-Inferiority — The overall non-inferiority was demonstrated if the lower limit of the 2-sided 95% CI was >-10% for all 4 serogroups. 95% CI of the difference was calculated from the Wilson Score method without continuity correction; Difference in Percentage of Participants = 8.75, 95% CI 2-sided [4.80 to 13.60]
Statistical Analysis 3: Comparison: Group 1a:MenACYW Conjugate Vaccine (Post 12-month Vaccination) vs Group 2a: MENVEO (Post 12-month Vaccination); Statistical analysis for Serogroup Y; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 2]; Difference in Percentage of Participants = 4.09, 95% CI 2-sided [0.68 to 8.44]
Statistical Analysis 4: Comparison: Group 1a:MenACYW Conjugate Vaccine (Post 12-month Vaccination) vs Group 2a: MENVEO (Post 12-month Vaccination); Statistical analysis for Serogroup W; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 2]; Difference in Percentage of Participants = 1.19, 95% CI 2-sided [-1.18 to 4.45]

2. Primary Outcome: Groups 1 and 2: Percentage of Participants Who Achieved Antibody Titers >=1:8 by hSBA at Day 30 Post 6-Month Vaccination
Description: Functional meningococcal antibody activity against serogroups A, C, Y, and W were measured in a serum bactericidal assay utilizing the hSBA. Percentages are rounded off to the tenth decimal place.
Time Frame: Day 30 post 6-month vaccination (Month 7)
Population: PPAS1 (for infant vaccination). PPAS1 included participants of FAS1 (subset of all randomized participants who received >=1 dose of the study vaccine in infancy [<12 months of age] and had a valid post-vaccination serology result in infancy) with no relevant protocol deviations during infancy. Only those participants with data collected for each specific serogroup are reported.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: MenACYW Conjugate Vaccine | Group 2: MENVEO
Number analyzed (Participants) | 883 | 438
percentage of participants
  Serogroup A: number analyzed (Participants) | 852 | 409
  Serogroup A | 77.9 [75.0 to 80.7] | 67.7 [63.0 to 72.2]
  Serogroup C: number analyzed (Participants) | 835 | 421
  Serogroup C | 99.0 [98.1 to 99.6] | 91.2 [88.1 to 93.7]
  Serogroup Y: number analyzed (Participants) | 861 | 423
  Serogroup Y | 98.3 [97.1 to 99.0] | 91.7 [88.7 to 94.2]
  Serogroup W | 98.6 [97.6 to 99.3] | 92.9 [90.1 to 95.1]
Statistical Analysis 1: Comparison: Group 1: MenACYW Conjugate Vaccine vs Group 2: MENVEO; Statistical analysis for Serogroup A; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 2]; Difference in Percentage of Participants = 10.21, 95% CI 2-sided [4.98 to 15.59]
Statistical Analysis 2: Comparison: Group 1: MenACYW Conjugate Vaccine vs Group 2: MENVEO; Statistical analysis for Serogroup C; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 2]; Difference in Percentage of Participants = 7.83, 95% CI 2-sided [5.31 to 10.96]
Statistical Analysis 3: Comparison: Group 1: MenACYW Conjugate Vaccine vs Group 2: MENVEO; Statistical analysis for Serogroup Y; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 2]; Difference in Percentage of Participants = 6.53, 95% CI 2-sided [4.01 to 9.62]
Statistical Analysis 4: Comparison: Group 1: MenACYW Conjugate Vaccine vs Group 2: MENVEO; Statistical analysis for Serogroup W; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 2]; Difference in Percentage of Participants = 5.72, 95% CI 2-sided [3.44 to 8.57]

3. Secondary Outcome: Groups 1 and 2: Percentage of Participants Who Achieved Anti-Hepatitis B Antibody Concentrations >=10 Milli-International Units Per Milliliter (mIU/mL) at Day 30 Post 6-Month Vaccination
Description: Anti-Hepatitis B surface antibodies (HBsAg) were measured by the commercially available VITROS ECi/ECiQ immunodiagnostic system using chemiluminescence detection technology. The percentage of participants with an anti-HBsAg antibody titer >=10 mIU/mL was assessed. Percentages are rounded off to the tenth decimal place.
Time Frame: Day 30 post 6-month vaccination (Month 7)
Population: Analysis was performed on PPAS1 (for infant vaccination) which included participants of FAS1 with no relevant protocol deviations during infancy. Only those participants with data collected are reported.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: MenACYW Conjugate Vaccine | Group 2: MENVEO
Number analyzed (Participants) | 765 | 348
percentage of participants | 98.6 (97.4) [97.4 to 99.3] | 98.0 (95.9) [95.9 to 99.2]

4. Secondary Outcome: Groups 1 and 2: Percentage of Participants Who Achieved Anti-Polyribosyl-Ribitol (PRP) Antibody Concentrations >=0.15 and >=1.0 Microgram (mcg)/mL at Day 30 Post 6-Month Vaccination
Description: Anti-PRP concentrations were measured using a farr-type radioimmunoassay (RIA). The percentage of participants with an PRP antibody titer >=0.15 mcg/mL and >=1.0 mcg/mL were assessed. Percentages are rounded off to the tenth decimal place.
Time Frame: Day 30 post 6-month vaccination (Month 7)
Population: Analysis was performed on PPAS1 (for infant vaccination) which included participants of FAS1 with no relevant protocol deviations during infancy. Only those participants with data collected for each specified category are reported.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: MenACYW Conjugate Vaccine | Group 2: MENVEO
Number analyzed (Participants) | 882 | 420
percentage of participants
  >=0.15 mcg/mL | 99.0 (98.1) [98.1 to 99.5] | 96.4 (94.2) [94.2 to 98.0]
  >=1.0 mcg/mL | 91.3 (89.2) [89.2 to 93.0] | 85.7 (82.0) [82.0 to 88.9]

5. Secondary Outcome: Groups 1 and 2: Percentage of Participants Who Achieved Anti-Poliovirus Antibody Titers >=1:8 at Day 30 Post 6-Month Vaccination
Description: Anti-poliovirus types 1, 2, and 3 were measured by neutralization assay. The percentage of participants with anti-polio antibody titers >=1:8 were assessed.
Time Frame: Day 30 post 6-month vaccination (Month 7)
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: MenACYW Conjugate Vaccine | Group 2: MENVEO
Number analyzed (Participants) | 854 | 415
percentage of participants
  Anti-polio 1: number analyzed (Participants) | 839 | 412
  Anti-polio 1 | 100 [99.6 to 100] | 100 [99.1 to 100]
  Anti-polio 2: number analyzed (Participants) | 838 | 406
  Anti-polio 2 | 100 [99.6 to 100] | 100 [99.1 to 100]
  Anti-polio 3 | 100 [99.6 to 100] | 100 [99.1 to 100]

6. Secondary Outcome: Groups 1 and 2: Percentage of Participants Who Achieved Anti-Rotavirus Immunoglobulin A (IgA) Antibody Concentrations >=3-Fold Rise at Day 30 Post 6-Month Vaccination
Description: Anti-rotavirus IgA antibodies in human serum were measured by enzyme-linked immunosorbent assay (ELISA). The percentage of participants who achieved anti-rotavirus IgA Ab concentrations >=3-fold rise were assessed. Percentages are rounded off to the tenth decimal place.
Time Frame: Day 30 post 6-month vaccination (Month 7)
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: MenACYW Conjugate Vaccine | Group 2: MENVEO
Number analyzed (Participants) | 663 | 321
percentage of participants | 91.0 (88.5) [88.5 to 93.0] | 92.8 (89.4) [89.4 to 95.4]

7. Secondary Outcome: Groups 1 and 2: Geometric Mean Concentrations (GMCs) of Anti-Rotavirus IgA Antibodies at Day 30 Post 6-Month Vaccination
Description: GMCs of anti-rotavirus serum IgA antibodies were assessed using ELISA.
Time Frame: Day 30 post 6-month vaccination (Month 7)
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: Units/mL
Arm/Group | Group 1: MenACYW Conjugate Vaccine | Group 2: MENVEO
Number analyzed (Participants) | 857 | 403
Units/mL | 272 (244) [244 to 303] | 308 (264) [264 to 360]

8. Secondary Outcome: Groups 1 and 2: GMCs of Anti-Pertussis Antibodies at Day 30 Post 6-Month Vaccination
Description: GMCs of anti-pertussis antibodies (pertussis toxoid [PT], filamentous hemagglutinin adhesin [FHA], pertactin [PRN] and fimbriae types 2 and 3 [FIM]) were measured by electrochemiluminescent (ECL) assay.
Time Frame: Day 30 post 6-month vaccination (Month 7)
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: ELISA units/mL
Arm/Group | Group 1: MenACYW Conjugate Vaccine | Group 2: MENVEO
Number analyzed (Participants) | 906 | 444
ELISA units/mL
  Anti-PT | 75.8 (72.2) [72.2 to 79.6] | 78.6 (72.8) [72.8 to 84.9]
  Anti-FHA | 95.7 (90.9) [90.9 to 101] | 98.6 (91.7) [91.7 to 106]
  Anti-PRN | 39.4 (36.8) [36.8 to 42.3] | 42.1 (37.9) [37.9 to 46.6]
  Anti-FIM | 309 (291) [291 to 330] | 311 (284) [284 to 341]

9. Secondary Outcome: Groups 1 and 2: GMCs of Anti-Pneumococcal Antibodies at Day 30 Post 6-Month Vaccination
Description: GMCs of anti-pneumococcal antibodies was assessed by pneumococcal capsular polysaccharide (PnPS) IgG ECL assay which is used to quantitate the amount of anti-streptococcus pneumoniae PS (serotypes 1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F and 23F) antibodies in human serum.
Time Frame: Day 30 post 6-month vaccination (Month 7)
Population: Analysis was performed on PPAS1 (for infant vaccination) which included participants of FAS1 with no relevant protocol deviations during infancy. Only those participants with data collected for each specified serotype are reported.
Measure: Geometric Mean (95% Confidence Interval); unit: mcg/mL
Arm/Group | Group 1: MenACYW Conjugate Vaccine | Group 2: MENVEO
Number analyzed (Participants) | 874 | 420
mcg/mL
  Serotype 1: number analyzed (Participants) | 872 | 420
  Serotype 1 | 2.26 [2.13 to 2.40] | 1.93 [1.77 to 2.12]
  Serotype 3: number analyzed (Participants) | 869 | 412
  Serotype 3 | 0.607 [0.577 to 0.638] | 0.544 [0.505 to 0.585]
  Serotype 4: number analyzed (Participants) | 872 | 420
  Serotype 4 | 1.46 [1.40 to 1.53] | 1.33 [1.24 to 1.42]
  Serotype 5: number analyzed (Participants) | 873 | 420
  Serotype 5 | 1.54 [1.46 to 1.63] | 1.26 [1.15 to 1.37]
  Serotype 6A | 4.01 [3.82 to 4.22] | 3.34 [3.09 to 3.62]
  Serotype 6B | 2.47 [2.29 to 2.67] | 1.97 [1.75 to 2.21]
  Serotype 7F: number analyzed (Participants) | 874 | 419
  Serotype 7F | 3.48 [3.32 to 3.64] | 3.40 [3.18 to 3.63]
  Serotype 9V: number analyzed (Participants) | 873 | 420
  Serotype 9V | 1.88 [1.78 to 1.99] | 1.61 [1.48 to 1.74]
  Serotype 14: number analyzed (Participants) | 872 | 420
  Serotype 14 | 6.95 [6.53 to 7.41] | 7.17 [6.58 to 7.81]
  Serotype 18C | 1.95 [1.86 to 2.04] | 1.82 [1.69 to 1.96]
  Serotype 19A | 2.21 [2.10 to 2.32] | 2.00 [1.86 to 2.14]
  Serotype 19F | 3.36 [3.21 to 3.52] | 2.98 [2.77 to 3.21]
  Serotype 23F: number analyzed (Participants) | 872 | 420
  Serotype 23F | 1.59 [1.49 to 1.69] | 1.30 [1.18 to 1.44]

10. Secondary Outcome: Groups 1a and 2a: Percentage of Participants Who Achieved Vaccine Response for Measles, Mumps and Rubella (MMR) Antibodies at Day 30 Post 12-Month Vaccination
Description: Vaccine response against anti-measles and anti-rubella antibodies were measured by bulk IgG enzyme immunoassay and anti-mumps antibodies were assessed by ELISA. Percentage of participants with anti-measles, anti-mumps, anti-rubella antibody concentration that met the respective mentioned criterion are reported: measles: >=255 mIU/mL; mumps: >=10 antibody units per milliliter and rubella: >=10 IU/mL. Percentages are rounded off to the tenth decimal place.
Time Frame: Day 30 post 12-month vaccination (Month 13)
Population: Analysis was performed on PPAS3 (for 2nd year of life vaccination) which included participants of FAS3 with no relevant protocol deviations. Only those participants with data collected for each specified category are reported.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1a:MenACYW Conjugate Vaccine (Post 12-month Vaccination) | Group 2a: MENVEO (Post 12-month Vaccination)
Number analyzed (Participants) | 662 | 301
percentage of participants
  Anti-measles | 97.6 [96.1 to 98.6] | 97.3 [94.8 to 98.8]
  Anti-mumps: number analyzed (Participants) | 660 | 301
  Anti-mumps | 95.5 [93.6 to 96.9] | 97.7 [95.3 to 99.1]
  Anti-rubella | 97.9 [96.5 to 98.8] | 98.0 [95.7 to 99.3]

11. Secondary Outcome: Groups 1a and 2a: Percentage of Participants Who Achieved Vaccine Response for Varicella Antibodies at Day 30 Post 12-Month Vaccination
Description: Vaccine response against anti-varicella antibodies were measured by glycoprotein (gp) ELISA. Percentage of participants with anti-varicella antibody concentration >=5 antibody (Ab) gpELISA units/mL are reported. Percentages are rounded off to the tenth decimal place.
Time Frame: Day 30 post 12-month vaccination (Month 13)
Population: Analysis was performed on PPAS3 (for 2nd year of life vaccination) which included participants of FAS3 with no relevant protocol deviations. Only those participants with data collected are reported.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1a:MenACYW Conjugate Vaccine (Post 12-month Vaccination) | Group 2a: MENVEO (Post 12-month Vaccination)
Number analyzed (Participants) | 662 | 301
percentage of participants | 96.4 [94.7 to 97.7] | 94.7 [91.5 to 96.9]

12. Secondary Outcome: Groups 1a and 2a: GMCs of Anti-Pneumococcal Antibodies at Day 30 Post 12-Month Vaccination
Description: GMCs of anti-pneumococcal antibodies was assessed by PnPS IgG ECL assay which is used to quantitate the amount of anti-streptococcus pneumoniae PS (serotypes 1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F and 23F) antibodies in human serum.
Time Frame: Day 30 post 12-month vaccination (Month 13)
Population: Analysis was performed on PPAS3 (for 2nd year of life vaccination) which included participants of FAS3 with no relevant protocol deviations. Only those participants with data collected for each specified serotype are reported.
Measure: Geometric Mean (95% Confidence Interval); unit: mcg/mL
Arm/Group | Group 1a:MenACYW Conjugate Vaccine (Post 12-month Vaccination) | Group 2a: MENVEO (Post 12-month Vaccination)
Number analyzed (Participants) | 653 | 300
mcg/mL
  Serotype 1: number analyzed (Participants) | 652 | 299
  Serotype 1 | 3.81 [3.56 to 4.08] | 3.44 [3.12 to 3.81]
  Serotype 3: number analyzed (Participants) | 651 | 299
  Serotype 3 | 0.771 [0.728 to 0.817] | 0.751 [0.690 to 0.818]
  Serotype 4: number analyzed (Participants) | 652 | 299
  Serotype 4 | 2.08 [1.95 to 2.22] | 2.00 [1.83 to 2.18]
  Serotype 5: number analyzed (Participants) | 652 | 300
  Serotype 5 | 2.70 [2.53 to 2.88] | 2.46 [2.25 to 2.69]
  Serotype 6A: number analyzed (Participants) | 652 | 300
  Serotype 6A | 9.65 [9.09 to 10.2] | 9.51 [8.72 to 10.4]
  Serotype 6B: number analyzed (Participants) | 649 | 300
  Serotype 6B | 7.41 [6.92 to 7.93] | 6.37 [5.77 to 7.03]
  Serotype 7F: number analyzed (Participants) | 652 | 298
  Serotype 7F | 5.40 [5.08 to 5.73] | 6.04 [5.56 to 6.55]
  Serotype 9V: number analyzed (Participants) | 652 | 299
  Serotype 9V | 3.53 [3.31 to 3.77] | 3.62 [3.30 to 3.96]
  Serotype 14 | 7.80 [7.26 to 8.38] | 9.20 [8.37 to 10.1]
  Serotype 18C: number analyzed (Participants) | 652 | 300
  Serotype 18C | 2.60 [2.44 to 2.78] | 2.92 [2.68 to 3.19]
  Serotype 19A: number analyzed (Participants) | 649 | 300
  Serotype 19A | 6.19 [5.82 to 6.59] | 5.86 [5.32 to 6.45]
  Serotype 19F: number analyzed (Participants) | 652 | 300
  Serotype 19F | 6.49 [6.11 to 6.90] | 6.01 [5.45 to 6.62]
  Serotype 23F: number analyzed (Participants) | 652 | 300
  Serotype 23F | 3.88 [3.60 to 4.17] | 3.41 [3.09 to 3.78]

13. Secondary Outcome: Groups 1b and 2b: Percentage of Participants Who Achieved Anti-PRP Antibody Concentrations >=1.0 mcg/mL at Day 30 Post 15-Month Vaccination
Description: Anti-PRP concentrations were measured using a farr-type RIA. The percentage of participants with an PRP antibody titers >=1.0 mcg/mL were assessed. Percentages are rounded off to the tenth decimal place.
Time Frame: Day 30 post 15-month vaccination (Month 16)
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Group 1b:MenACYW Conjugate Vaccine(Post 15-month Vaccination): Participants received MenACYW conjugate vaccine at 2, 4, 6, and 15 to 18 months of age and routine vaccines at 2, 4, 6, 12 to 15 and 15 to 18 months of age. The time of analyses as well as the collection of blood samples conducted in the 2nd year of life for this subgroup was 30 days after the 15-month vaccination.
- Group 2b: MENVEO (Post 15- Month Vaccination): Participants received MENVEO at 2, 4, 6, and 12 months of age and routine vaccines at 2, 4, 6, 12, and 15 to 18 months of age. The time of analyses as well as the collection of blood samples conducted in the 2nd year of life for this subgroup was 30 days after the 15-month vaccination.
Arm/Group | Group 1b:MenACYW Conjugate Vaccine(Post 15-month Vaccination) | Group 2b: MENVEO (Post 15- Month Vaccination)
Number analyzed (Participants) | 297 | 125
percentage of participants | 98.3 [96.1 to 99.5] | 98.4 [94.3 to 99.8]

14. Secondary Outcome: Groups 1b and 2b: Percentage of Participants Who Achieved Anti-Poliovirus Antibody Titers >=1:8 at Day 30 Post 15-Month Vaccination
Description: Anti-poliovirus types 1, 2, and 3 were measured by neutralization assay. The percentage of participants with anti-polio antibody titers >=1:8 are assessed.
Time Frame: Day 30 post 15-month vaccination (Month 16)
Population: as for outcome 10
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1b:MenACYW Conjugate Vaccine(Post 15-month Vaccination) | Group 2b: MENVEO (Post 15- Month Vaccination)
Number analyzed (Participants) | 291 | 122
percentage of participants
  Anti-polio 1: number analyzed (Participants) | 286 | 122
  Anti-polio 1 | 100 [98.7 to 100] | 100 [97.0 to 100]
  Anti-polio 2 | 100 [98.7 to 100] | 100 [97.0 to 100]
  Anti-polio 3: number analyzed (Participants) | 289 | 122
  Anti-polio 3 | 100 [98.7 to 100] | 100 [97.0 to 100]

15. Secondary Outcome: Groups 1b and 2b: Percentage of Participants Who Achieved Vaccine Response for Anti-Pertussis Antibodies at Day 30 Post 15-Month Vaccination
Description: Vaccine response was defined as: if the pre-booster (4th) vaccination concentration was <lower limit of quantification (LLOQ), then the post-booster (4th) vaccination concentration should be >=4 times LLOQ. The LLOQ was equal to 2.00 EU/mL. Percentages are rounded off to the tenth decimal place.
Time Frame: Day 30 post 15-month vaccination (Month 16)
Population: as for outcome 10
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1b:MenACYW Conjugate Vaccine(Post 15-month Vaccination) | Group 2b: MENVEO (Post 15- Month Vaccination)
Number analyzed (Participants) | 273 | 121
percentage of participants
  Anti-PT | 98.5 [96.3 to 99.6] | 98.3 [94.2 to 99.8]
  Anti-FHA | 96.7 [93.8 to 98.5] | 96.7 [91.8 to 99.1]
  Anti-PRN | 96.3 [93.4 to 98.2] | 97.5 [92.9 to 99.5]
  Anti-FIM | 98.2 [95.8 to 99.4] | 97.5 [92.9 to 99.5]

16. Secondary Outcome: Groups 1a and 2a: Geometric Mean Titers (GMTs) of Antibodies Against Meningococcal Serogroups A, C, Y, and W Measured by hSBA at Day 30 Post 6-Month Vaccination and Day 0 Before 12-Month Vaccination
Description: GMTs of antibody against meningococcal serogroups A, C, Y, and W were measured by hSBA. PPAS2 included participants of FAS2 (subset of all randomized participants who received >=1 dose of the study vaccine in infancy [at Visit 1 to 3, < 12 months of age] and had a valid pre-vaccination serology result at Visit 5 before the 12-month vaccinations for Subgroups 1a and 2a or at Visit 6 before the 15-month vaccinations for Subgroups 1b and 2b) with no relevant protocol deviations during infancy and for whom a pre-dose serology sample at Visit 5 for Subgroups 1a and 2a before the 12-month vaccinations or Visit 6 for Subgroups 1b and 2b before the 15-month vaccinations was not withdrawn.
Time Frame: Day 30 post 6-month vaccination (Month 7) and Day 0 before 12-month vaccination (Month 12)
Population: Analysis was performed on PPAS2 (for immunogenicity persistence evaluation). Only those participants with data collected for each specified category are reported. 3rd dose is 6-month vaccination and 4th dose is 12-month vaccination.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Groups:
- Group 2a: MENVEO (Post 12- Month Vaccination): Participants received MENVEO at 2, 4, 6, and 12 months of age and routine vaccines at 2, 4, 6, 12, and 15 to 18 months of age. The time of analyses as well as the collection of blood samples conducted in the 2nd year of life for this subgroup was 30 days after the 12-month vaccination.
Arm/Group | Group 1a:MenACYW Conjugate Vaccine (Post 12-month Vaccination) | Group 2a: MENVEO (Post 12- Month Vaccination)
Number analyzed (Participants) | 644 | 329
titer
  Serogroup A: Day 30 post 3rd dose: number analyzed (Participants) | 547 | 258
  Serogroup A: Day 30 post 3rd dose | 24.9 [21.6 to 28.6] | 16.3 [13.5 to 19.6]
  Serogroup A: Day 0 before 4th dose: number analyzed (Participants) | 627 | 321
  Serogroup A: Day 0 before 4th dose | 9.33 [8.45 to 10.3] | 6.43 [5.64 to 7.33]
  Serogroup C: Day 30 post 3rd dose: number analyzed (Participants) | 542 | 268
  Serogroup C: Day 30 post 3rd dose | 365 [325 to 411] | 51.4 [42.9 to 61.5]
  Serogroup C: Day 0 before 4th dose: number analyzed (Participants) | 637 | 324
  Serogroup C: Day 0 before 4th dose | 57.8 [51.5 to 64.8] | 4.82 [4.22 to 5.50]
  Serogroup Y: Day 30 post 3rd dose: number analyzed (Participants) | 558 | 270
  Serogroup Y: Day 30 post 3rd dose | 83.0 [75.0 to 91.8] | 42.9 [36.7 to 50.0]
  Serogroup Y: Day 0 before 4th dose: number analyzed (Participants) | 633 | 327
  Serogroup Y: Day 0 before 4th dose | 42.9 [39.3 to 46.7] | 10.4 [9.15 to 11.9]
  Serogroup W: Day 30 post 3rd dose: number analyzed (Participants) | 571 | 277
  Serogroup W: Day 30 post 3rd dose | 92.8 [84.8 to 102] | 51.4 [43.9 to 60.0]
  Serogroup W: Day 0 before 4th dose | 57.8 [52.7 to 63.3] | 9.27 [8.15 to 10.5]

17. Secondary Outcome: Groups 1a and 2a: Percentage of Participants Who Achieved Antibody Titers >=1:4 and >=1:8 Against Meningococcal Serogroups A, C, Y, and W at Day 30 Post 6-Month Vaccination and Day 0 Before 12-Month Vaccination
Description: Antibody titers of Meningococcal Serogroups A, C, Y, and W were measured by hSBA assay. PPAS2 included participants of FAS2 with no relevant protocol deviations during infancy and for whom a pre-dose serology sample at Visit 5 for Subgroups 1a and 2a before the 12-month vaccinations or Visit 6 for Subgroups 1b and 2b before the 15-month vaccinations was not withdrawn. Percentages are rounded off to the tenth decimal place.
Time Frame: Day 30 post 6-month vaccination (Month 7) and Day 0 before 12-month vaccination (Month 12)
Population: Analysis was performed on PPAS2 (for immunogenicity persistence evaluation). Only those participants with data collected for each specified category are reported. 3rd dose is 6-month vaccination, 4th dose is 12-month vaccination. D0 is Day 0 and D30 is Day 30.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1a:MenACYW Conjugate Vaccine (Post 12-month Vaccination) | Group 2a: MENVEO (Post 12- Month Vaccination)
Number analyzed (Participants) | 644 | 329
percentage of participants
  Serogroup A: D30 post 3rd dose:>=1:4: number analyzed (Participants) | 547 | 258
  Serogroup A: D30 post 3rd dose:>=1:4 | 87.0 [83.9 to 89.7] | 84.9 [79.9 to 89.0]
  Serogroup A: D30 post 3rd dose:>=1:8: number analyzed (Participants) | 547 | 258
  Serogroup A: D30 post 3rd dose:>=1:8 | 77.3 [73.6 to 80.8] | 70.2 [64.2 to 75.7]
  Serogroup A:D0 before 4th dose:>=1:4: number analyzed (Participants) | 627 | 321
  Serogroup A:D0 before 4th dose:>=1:4 | 82.5 [79.2 to 85.4] | 66.4 [60.9 to 71.5]
  Serogroup A:D0 before 4th dose:>=1:8: number analyzed (Participants) | 627 | 321
  Serogroup A:D0 before 4th dose:>=1:8 | 59.0 [55.0 to 62.9] | 47.0 [41.5 to 52.7]
  Serogroup C: D30 post 3rd dose:>=1:4 (n=): number analyzed (Participants) | 542 | 268
  Serogroup C: D30 post 3rd dose:>=1:4 (n=) | 99.3 [98.1 to 99.8] | 93.7 [90.0 to 96.3]
  Serogroup C: D30 post 3rd dose:>=1:8: number analyzed (Participants) | 542 | 268
  Serogroup C: D30 post 3rd dose:>=1:8 | 99.1 [97.9 to 99.7] | 91.0 [87.0 to 94.2]
  Serogroup C:D0 before 4th dose:>=1:4: number analyzed (Participants) | 637 | 324
  Serogroup C:D0 before 4th dose:>=1:4 | 95.4 [93.5 to 96.9] | 49.1 [43.5 to 54.7]
  Serogroup C:D0 before 4th dose:>=1:8: number analyzed (Participants) | 637 | 324
  Serogroup C:D0 before 4th dose:>=1:8 | 92.9 [90.7 to 94.8] | 34.0 [28.8 to 39.4]
  Serogroup Y: D30 post 3rd dose:>=1:4: number analyzed (Participants) | 558 | 270
  Serogroup Y: D30 post 3rd dose:>=1:4 | 99.1 [97.9 to 99.7] | 96.3 [93.3 to 98.2]
  Serogroup Y: D30 post 3rd dose:>=1:8: number analyzed (Participants) | 558 | 270
  Serogroup Y: D30 post 3rd dose:>=1:8 | 98.6 [97.2 to 99.4] | 92.2 [88.4 to 95.1]
  Serogroup Y:D0 before 4th dose:>=1:4: number analyzed (Participants) | 633 | 327
  Serogroup Y:D0 before 4th dose:>=1:4 | 99.2 [98.2 to 99.7] | 83.5 [79.0 to 87.3]
  Serogroup Y:D0 before 4th dose:>=1:8: number analyzed (Participants) | 633 | 327
  Serogroup Y:D0 before 4th dose:>=1:8 | 96.8 [95.2 to 98.1] | 69.1 [63.8 to 74.1]
  Serogroup W: D30 post 3rd dose:>=1:4: number analyzed (Participants) | 571 | 277
  Serogroup W: D30 post 3rd dose:>=1:4 | 99.8 [99.0 to 100] | 97.5 [94.9 to 99.0]
  Serogroup W: D30 post 3rd dose:>=1:8: number analyzed (Participants) | 571 | 277
  Serogroup W: D30 post 3rd dose:>=1:8 | 98.8 [97.5 to 99.5] | 94.2 [90.8 to 96.7]
  Serogroup W:D0 before 4th dose:>=1:4 | 98.9 [97.8 to 99.6] | 82.7 [78.1 to 86.6]
  Serogroup W:D0 before 4th dose:>=1:8 | 97.2 [95.6 to 98.3] | 62.0 [56.5 to 67.3]

ADVERSE EVENTS:
Time Frame: From first administration of study treatment (Day 0) up to 6-months post last administration of study treatment, approximately 24 months for Group 1 and 18 months for Group 2.
Description: Analysis was performed on safety analysis set which was defined as those participants who received at least 1 dose of the study vaccines and had any safety data available. All participants had safety analyzed according to the vaccine received post first dose.
Arm/Group | Group 1: MenACYW Conjugate Vaccine | Group 2: MENVEO
All-Cause Mortality (participants affected / at risk) | 1/1727 | 0/867
Serious Adverse Events (participants affected / at risk) | 99/1727 | 38/867
Other Adverse Events (participants affected / at risk) | 1471/1727 | 746/867
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: MenACYW Conjugate Vaccine (N=1727) | Group 2: MENVEO (N=867)
Craniocerebral Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Femur Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Head Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post Vaccination Fever (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Skull Fracture (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Skull Fractured Base (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Subdural Haematoma (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Upper Limb Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Cardiac Arrest (Cardiac disorders) | 1 (1) | 0 (0)
Congenital Absence Of Bile Ducts (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Pyloric Stenosis (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Talipes (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Urachal Abnormality (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Coagulopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Epilepsy (Nervous system disorders) | 0 (0) | 1 (1)
Febrile Convulsion (Nervous system disorders) | 8 (11) | 3 (4)
Infantile Spasms (Nervous system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 3 (4) | 1 (1)
Seizure Like Phenomena (Nervous system disorders) | 1 (1) | 0 (0)
Subarachnoid Haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 2 (2) | 0 (0)
Sandifer's Syndrome (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (2) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 3 (3) | 4 (4)
Ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Type 1 Diabetes Mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Abscess Neck (Infections and infestations) | 0 (0) | 1 (1)
Adenovirus Infection (Infections and infestations) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Bacterial Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Bordetella Infection (Infections and infestations) | 1 (1) | 0 (0)
Bronchiolitis (Infections and infestations) | 15 (16) | 4 (4)
Covid-19 (Infections and infestations) | 1 (1) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Croup Infectious (Infections and infestations) | 2 (2) | 0 (0)
Eczema Coxsackium (Infections and infestations) | 1 (1) | 0 (0)
Escherichia Urinary Tract Infection (Infections and infestations) | 1 (1) | 0 (0)
Exanthema Subitum (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 2 (2) | 3 (3)
Gastroenteritis Norovirus (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis Viral (Infections and infestations) | 1 (1) | 0 (0)
Gastrointestinal Viral Infection (Infections and infestations) | 1 (1) | 0 (0)
Impetigo (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 4 (5) | 1 (1)
Otitis Media (Infections and infestations) | 1 (1) | 0 (0)
Otitis Media Acute (Infections and infestations) | 1 (1) | 1 (1)
Parainfluenzae Virus Infection (Infections and infestations) | 2 (3) | 0 (0)
Perirectal Abscess (Infections and infestations) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Pharyngitis Streptococcal (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 6 (6) | 2 (2)
Pneumonia Mycoplasmal (Infections and infestations) | 1 (1) | 1 (1)
Pneumonia Viral (Infections and infestations) | 2 (2) | 0 (0)
Pyelonephritis (Infections and infestations) | 3 (3) | 0 (0)
Pyelonephritis Acute (Infections and infestations) | 2 (2) | 0 (0)
Respiratory Syncytial Virus Bronchiolitis (Infections and infestations) | 9 (9) | 4 (4)
Respiratory Syncytial Virus Infection (Infections and infestations) | 7 (7) | 6 (6)
Rhinovirus Infection (Infections and infestations) | 1 (1) | 0 (0)
Roseola (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Skin Bacterial Infection (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal Scalded Skin Syndrome (Infections and infestations) | 0 (0) | 1 (1)
Systemic Infection (Infections and infestations) | 1 (1) | 0 (0)
Systemic Viral Infection (Infections and infestations) | 1 (1) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 2 (2) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 2 (2) | 3 (4)
Viral Infection (Infections and infestations) | 1 (1) | 1 (1)
Glioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Apnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (3)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: MenACYW Conjugate Vaccine (N=1727) | Group 2: MENVEO (N=867)
Somnolence (Nervous system disorders) | 975 (2319) | 507 (1273)
Teething (Gastrointestinal disorders) | 106 (124) | 62 (73)
Vomiting (Gastrointestinal disorders) | 417 (607) | 196 (276)
Decreased Appetite (Metabolism and nutrition disorders) | 704 (1246) | 388 (732)
Nasopharyngitis (Infections and infestations) | 96 (105) | 50 (62)
Otitis Media (Infections and infestations) | 79 (91) | 48 (64)
Upper Respiratory Tract Infection (Infections and infestations) | 214 (264) | 130 (162)
Crying (General disorders) | 1023 (2366) | 541 (1303)
Injection Site Bruising (General disorders) | 185 (380) | 88 (158)
Injection Site Erythema (General disorders) | 806 (3898) | 409 (2054)
Injection Site Pain (General disorders) | 1201 (9341) | 637 (5053)
Injection Site Swelling (General disorders) | 632 (2651) | 323 (1491)
Pyrexia (General disorders) | 580 (912) | 312 (512)
Irritability (Psychiatric disorders) | 1154 (3082) | 598 (1694)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications.

DOCUMENTS (2):
  • Study Protocol (2022-01-26): https://cdn.clinicaltrials.gov/large-docs/08/NCT03537508/Prot_000.pdf
  • Statistical Analysis Plan (2024-01-22): https://cdn.clinicaltrials.gov/large-docs/08/NCT03537508/SAP_001.pdf